CLINICAL TRIAL: NCT06740175
Title: The Feasibility of Multispectral Optoacoustic Tomography in Different Diseases: a Phase 1 Explorative Imaging Study (FOMO-study)
Brief Title: The Feasibility of Multispectral Optoacoustic Tomography in Different Diseases
Acronym: FOMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL71894.042.19
Record Dates: First submitted 2024-11-07; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Sjogren Syndrome; Malignant Tumors; Arterial Disease
Keywords: Multispectral optoacoustic tomography; Optoacoustic imaging; Sjogren syndrome; Diagnostic; Diagnose; Non-invasive
MeSH Terms: conditions — Sjogren's Syndrome; Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental MSOT measurement (Experimental): imaged with the multispectral optoacoustic tomography device (MSOT Acuity Echo).
  Interventions: Device: Multispectral optoacoustic tomography

INTERVENTIONS:
Device: Multispectral optoacoustic tomography — If patients are willing to participate in this study, they are imaged with the multispectral optoacoustic tomography device (MSOT Acuity Echo) at the department of nuclear medicine and molecular imaging. The imaging procedure takes 15 minutes at most.

SUMMARY:
Optoacoustic imaging is a new and innovative imaging technique that combines the high contrast of optical imaging with the penetration depth and high spatial resolution of ultrasonography using the optoacoustic effect. It can resolve different endogenous tissue chromophores and may thereby provide insight in molecular changes associated with disease (-progression). It can be potentially used as an technique for diagnosis, treatment monitoring and disease localization. As the technique is relatively new in the clinical setting, there is not much clinical experience with optoacoustic imaging. The rationale for this study is to assess the technical feasibility of optoacoustic imaging in a variety of disease and to determine endogenous biomarkers for disease characterization for potential diagnosis and/or disease monitoring.

DETAILED DESCRIPTION:
Optoacoustic imaging is a novel imaging method that is based on the optoacoustic effect, first described by Alexander Graham Bell in 1880. When biological tissue is illuminated with an ultrashort laser pulse, tissue chromophores absorb laser light and form pressure transient waves as a result of thermoelastic expansion. These optoacoustic or photoacoustic waves can be detected by wideband ultrasonic transducers around the tissue. Optoacoustic imaging is unique as it resolves optical contrast, but the resolution obeys the rules of ultrasonic diffraction; scattering of the ultrasonic signal in tissue is much weaker than for optical signals. Therefore, optoacoustic methods are insensitive to photon scattering within biological tissues and thereby provide higher spatial resolution with high sensitivity to tissue light absorption. In addition, it obtains penetration depths up to several centimeters, making it suitable for imaging deeper tissues within the body. Optoacoustic imaging has been shown to address clinically relevant aspects of various diseases, such as multiple prevalent cancers and inflammatory bowel disease.

Multiple imaging methods are based on optoacoustic imaging. However, unlike other types of optoacoustic imaging, multispectral optoacoustic tomography (MSOT) involves illumination of tissue with multiple wavelengths. Due to the high frequency pulse rate of the 9 laser, multiple wavelengths can be identified in one single image. Images can be processed using spectral unmixing algorithms in order to resolve different tissue chromophores, such as hemoglobin, deoxyhemoglobin, melanin and fat, which all have a distinct absorption spectrum or "spectral signature". This provides the ability to reconstruct an image by distinguishing and quantifying the contribution of specific absorbers including endogenous tissue chromophores.

Differences in the distribution of endogenous chromophores between normal tissue and diseased-tissue have been described extensively in preclinical and clinical optoacoustic studies. As the proliferation and metastatic spread in malignant tumors is highly dependent on angiogenesis, differences in hemoglobin concentration between normal tissue and tumor tissue is a well-known pathophysiological phenomenon Abnormal vascularization causing a local increase in hemoglobin concentration produces strong optoacoustic contrast, making optoacoustic imaging suitable for visualization of angiogenesis and tumors. This phenomenon could be used for diagnosis of a variety of malignant tumors, but potentially also for monitoring of disease progression after treatment. For example, relevant differences between hemoglobin distribution in benign and malignant thyroid tissue have been observed and the visualization of breast tumors using otoacoustics has been described.

For peripheral arterial disease, hemoglobin distribution and plaque characteristics are highly relevant biological features in the characterization of the disease. Nowadays, imaging modalities like X-ray CT are considered the gold standard, which give a relevant radiation burden to patients. Optoacoustic imaging has the potential for visualizing for example the peripheral arteries and the carotid artery, even in a 3D setting Identification of specific plaque characteristics like collagen and lipids would be a next step forward in visualization of plaque biology and its relationship with plaque rupture. This is topic of an already approved MSOT protocol in which 5 patients are enrolled.

As MSOT is experiencing a surge of interest in clinical investigation, there have been technological developments that enable imaging systems suitable for clinical use. The MSOT Acuity Echo (iThera Medical GmbH) that we use in the UMCG is dedicated for clinical research and similar to clinical ultra-sound technology in form and handling. Furthermore, it enables additional use of ultrasonography (OPUS) so that it delivers anatomical, functional and molecular information simultaneously. The MSOT Acuity Echo provides immediate feedback in the form of live images.

As multiple disciplines (surgery, radiology, nuclear medicine, oral and maxillofacial surgery, internal medicine) are interested in using the device, we aim to explore the possibilities of MSOT for various indications. We hypothesize that visualizing tissue chromophores with MSOT can lead to identification of molecular changes associated with disease (-progression).

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diseases will be included:

  1. Morbus Sjögren,
  2. A superficially located malignant tumor < 5 centimeter beneath the skin
  3. (Peripheral) arterial disease
* Age ≥ 18 years;

Exclusion Criteria:

* Patients with disease localizations or manifestations that do not enable good coupling between the optoacoustic probe and the skin, as decided by the researchers;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Pregnant women. Women of childbearing potential need to undergo a pregnancy test before participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Optoacoustic Signal Analysis | After informed consent the patient will be imaged for 15 minutes.
  Quantitative assessment of optoacoustic signals from tissue chormophores (e.g., hemoglobine, deoxyhemaglobine, water, lipid, and collagen). The signal of the different chormophores are described as arbitrary units (a.u.)
Comparison with Standard Imaging Modalities | After informed consent the patient will be imaged for 15 minutes.
  Validation of optoacoustic imaging by comparing chromophore signals to imaging features from CT, MRI, PET, and/or ultrasound. Correlation coefficients or diagnostic accuracy metrics (e.g., sensitivity, specificity, area under the curve).
Histopathological Correlation | After informed consent the patient will be imaged for 15 minutes.
  Correlation of optoacoustic findings with histopathological results from biopsy or surgical specimens. Agreement rate or correlation metrics (e.g. p-values)

CONTACTS AND LOCATIONS:
Locations (1):
- University medical center groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Relevant research data on request
Supporting Information: Study Protocol, CSR
Time Frame: It will be available after the end date of the study. It will be available for 15 years after the study has ended
Access Criteria: PI and other researchers on request. They are able to access the Study Protocol and the Clinical Study Report